CLINICAL TRIAL: NCT02861560
Title: A Case Series to Investigate the Safety and Efficacy of Weekly Application of Dehydrated Human Amnion/Chorion Membrane (dHACM) in the Treatment of Pressure Ulcers
Brief Title: Case Series of Weekly Applications of dHACM in Treatment of Pressure Ulcers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MiMedx Group, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EFPU001
Record Dates: First submitted 2016-08-05; First posted 2016-08-10 (Estimated); Last update posted 2018-08-24 (Actual); Status verified 2018-08

CONDITIONS: Pressure Ulcer
MeSH Terms: conditions — Pressure Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- dHACM (Experimental): Dehydrated human amnion/chorion membrane (dHACM)
  Interventions: Other: dHACM

INTERVENTIONS:
Other: dHACM — Dehydrated human amnion/chorion membrane (dHACM) product and is regulated as a Human Cells, Tissues and Cellular and Tissue Based Product (HCT/P) under Section 361 of the Public Health Service Act by the Food and Drug Administration (FDA)

SUMMARY:
A prospective case series investigating the efficacy and safety of dehydrated human amnion/chorion membrane (dHACM) in the treatment of patients with Stage II or III pressure ulcers

ELIGIBILITY:
Inclusion Criteria:

1. Index ulcer characteristics:

   1. Ulcer present for ≥ 30 days (Day 0)
   2. Index ulcer is located spine, lower back or buttocks
   3. Index ulcer area after debridement is ≥ 2 cm² and ≤ 25 cm² at the randomization visit
   4. Ulcer must be Stage II or III as determined by the National Pressure Ulcer Advisory Panel (NPUAP) pressure ulcer staging system
2. Subject criteria must include:

   1. Age 16 or older
   2. The subject is willing and able to provide informed consent and participate in all procedures and follow-up evaluations necessary to complete the study (minors will provide assent with consent provided by parent)

Exclusion Criteria:

1. Index ulcer characteristics that will make subject ineligible for enrollment:

   1. Stage I or IV ulcers as determined by NPUAP pressure ulcer staging system
   2. Signs and symptoms of local infection
   3. Previous surgical procedure performed at site
   4. Known or suspected local skin malignancy at index ulcer site
   5. Prior radiation therapy treatment at the index ulcer site
2. Subject criteria that will make subject ineligible for enrollment:

   1. Presence of other diseases which, in the Opinion of the Investigator, may result in allograft failure or has experienced graft failure in the past (examples include: immune system disorders including Systemic Lupus Erythematosus (SLE), Fibromyalgia, Acquired Immunodeficiency Syndrome (AIDS) or HIV)
   2. Currently taking medications which in the opinion of the investigator may affect graft incorporation
   3. Allergy or known sensitivity to Aminoglycosides such as gentamicin sulfate and/or streptomycin sulfate
   4. Any condition(s) that in the opinion of the investigator may seriously compromises the subject's ability to participate in this study. Examples include: known history of poor adherence with medical treatment, current drug or alcohol abuse or a medical/psychiatric condition
   5. Pregnancy at enrollment or within last 6 months, women who are breastfeeding, or women of childbearing potential who are planning to become pregnant during the time of the study OR are unwilling/unable to use acceptable methods of contraception (birth control pills, barriers, or abstinence)
   6. Subjects currently enrolled in this study (i.e. concurrent enrollment in the study is prohibited)
   7. Subject has used any investigational drug(s) or therapeutic device(s) within 30 days preceding screening.
   8. Any pathology that would limit the blood supply and compromise healing
   9. Subject is a prisoner

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2016-05; Primary Completion 2018-05 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
Healing Rate | 8 weeks

SECONDARY OUTCOMES:
Adverse Events | 8 Weeks
Quality of Life | 8 Weeks
  SF-36 Health Survey

CONTACTS AND LOCATIONS:
Overall Officials: Donald Fetterolf, MD, Study Director — Chief Medical Officer
Locations (1):
- Shepherd Spine Center, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No